CLINICAL TRIAL: NCT05721937
Title: CIBINQO™ Pregnancy Registry: An Observational Study of the Safety of Abrocitinib Exposure in Pregnant Women and Their Offspring
Brief Title: A Study of How Safe Abrocitinib (CIBINQO) is in Pregnant Women and Their Offspring
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451095; NCT05721937 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-01-26; First posted 2023-02-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: pregnancy; dermatitis, atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Exposed to CIBINQO during pregnancy: Received at least one dose of CIBINQO at any time during pregnancy or prior to pregnancy (within 1 day prior to the date of conception).
  Interventions: Drug: Abrocitinib
- Unexposed to CIBINQO during pregnancy: Diagnosed with moderate-to-severe atopic dermatitis, but not exposed to CIBINQO during pregnancy.

INTERVENTIONS:
Drug: Abrocitinib — taken by mouth
  Groups: Exposed to CIBINQO during pregnancy

SUMMARY:
The purpose of this observational study is to learn about the safety of abrocitinib (CIBINQO) in pregnant women and the offspring.

The study is seeking participants who:

* Are currently or recently pregnant
* Receive at least one dose of CIBINQO at any time during pregnancy or prior to pregnancy OR have a diagnosis of moderate-to-severe atopic dermatitis

All participants in this study will receive treatment according to routine care, as this is an observational study. The exposed group will consist of pregnant women exposed to abrocitinib during pregnancy. The unexposed group will consistent of pregnant women with moderate-to-severe atopic dermatitis who are not exposed to abrocitinib during pregnancy.

The study will compare the experiences of pregnant women receiving abrocitinib to pregnant women who do not. This will help us determine if abrocitinib is safe during pregnancy.

Participants will take part in this study until their infant is 12 months of age. During this time, the participant's care will be managed no differently than if she was not taking part in this study. Data will be collected through a virtual research coordinating center at enrollment, the end of the second trimester, and pregnancy outcome (live birth or fetal loss). For live-born infants, data on the infants will be collected at 4 and 12 months of age. No additional visits beyond routine care will be required.

ELIGIBILITY:
Inclusion Criteria:

* Women of any age who are currently or recently pregnant (recently pregnant defined as enrollment within 1 year of pregnancy outcome)
* Consent to participate in this study and evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study
* Authorization for her healthcare provider(s) to provide data to the registry
* Must receive at least one dose of CIBINQO at any time during pregnancy or prior to pregnancy (within 1 day prior to the date of conception) OR have a diagnosis of moderate-to-severe atopic dermatitis at any time prior to pregnancy outcome.

Exclusion Criteria:

* Participants will be excluded from the registry if they do not meet the inclusion criteria listed above.

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will include pregnant women of any age who meet the eligibility criteria for inclusion. The exposed cohort will include women who are exposed to CIBINQO at any time during pregnancy. All pregnant women exposed to CIBINQO will be eligible to participate in the registry, but the analysis population will be limited to women with moderate-to-severe AD. The primary comparator group will include women with moderate to- severe AD who are unexposed to CIBINQO during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent of live birth children with major congenital malformations | Enrollment until 12 months after delivery
  An abnormality of body structure or function that is present at birth, is of prenatal origin (i.e., birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention.

SECONDARY OUTCOMES:
Percent of participants with children with minor congenital malformations | Enrollment until 12 months after delivery
  An anomaly or abnormality of body structure that is present at birth, is of prenatal origin (i.e., birth defect), poses no significant health problem in the neonatal period, and tends to have limited social or cosmetic consequences for the affected individual.
Percent of participants with spontaneous abortion | Enrollment until end of pregnancy (up to 20 gestational weeks)
  An involuntary fetal loss or the expulsion of the products of conception occurring at <20 gestational weeks.
Percent of participants with stillbirths | Enrollment until end of pregnancy (up to 9 months)
  An involuntary fetal loss occurring at ≥20 gestational weeks or, if gestational age is unknown, a fetus weighing ≥350 g.
Percentage of participants with an elective termination | Enrollment until end of pregnancy (up to 9 months)
  A voluntary fetal loss or interruption of pregnancy that occurs for any reason, including but not limited to for the preservation of maternal health or due to fetal abnormalities
Percent of participants with preterm birth | Enrollment until 12 months after delivery
  A live birth occurring at <37 gestational weeks.
Percent of participants with children born small for gestational age | Enrollment until 12 months after delivery
  Birthweight <10th percentile for sex and gestational age using standard growth charts for full and preterm live born infants.
Percentage of participants with children with postnatal growth deficiency | Enrollment until 12 months after delivery
  Weight, length, or head circumference in <10th percentile for sex and chronological age using standard growth charts
Percent of participants with infant developmental delay | Enrollment until 12 months after delivery
  Failure to achieve the developmental milestones for chronological age, as defined by the CDC.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451095